CLINICAL TRIAL: NCT03307993
Title: Interventional, Open-label, Positron Emission Tomography (PET) Study Investigating the Brain Receptor Occupancy of Idalopirdine in Patients With Alzheimer's Disease
Brief Title: Positron Emission Tomography (PET) Study in Patients With Alzheimer's Disease
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated for strategic reasons.
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17475A
Record Dates: First submitted 2017-09-26; First posted 2017-10-12 (Actual); Last update posted 2018-04-04 (Actual); Status verified 2018-04

CONDITIONS: Alzheimer's Disease
Keywords: Lu AE58054
MeSH Terms: conditions — Alzheimer Disease | interventions — (2-(6-fluoro-1H-indol-3-yl)-ethyl)-(3-(2,2,3,3-tetrafluoropropoxy)benzyl)amine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Idalopirdine (Experimental): Idalopirdine 60 mg once daily for 10 day (up to 14 days possible), adjunct to donezepil (patients individualized maintenance dose)
  If high receptor occupancy cannot be verified, the receptor occupancy following a higher dose (up to 60 mg twice daily for 10-14 days) will be assessed in Cohort 2.
  Interventions: Drug: Idalopirdine

INTERVENTIONS:
Drug: Idalopirdine — Idalopirdine 60-120 mg daily dose
  Other Names: Lu AE58054

SUMMARY:
To investigate the brain receptor occupancy of idalopirdine in patients with Alzheimer's disease (AD)

ELIGIBILITY:
Inclusion Criteria:

* The patient has probable AD diagnosed according to National Institute of Neurological and Communicative Disorders and Stroke and the Alzheimer's disease and Related Disorders Association (NINCDS-ADRDA) criteria.
* The patient has had a positive amyloid PET scan, which in the opinion of the principal investigator is consistent with a diagnosis of AD.
* The patient has a Mini Mental State Examination (MMSE) score at screening of at least 15 and no greater than 22.
* The patient has a knowledgeable and reliable caregiver who will accompany the patient to all clinic visits during the study and answer questions about the patient.
* The patient is a man or woman of at least 50 years of age and has a body mass index (BMI) ≥ 18.5 kg/m2.

Exclusion Criteria:

* The patient has evidence of any clinically significant neurodegenerative disease, or other serious neurological disorders other than AD including but not limited to Lewy body dementia, fronto-temporal dementia, Parkinson's disease, Huntington's disease, major cortical stroke, major head trauma, primary or secondary cerebral neoplasia or systemic medical diseases that are, in the investigator's opinion, likely to affect central nervous system functioning and may influence the outcome or analysis of the scan results.
* The patient is, in the investigator's opinion, unlikely to comply with the protocol or is unsuitable for any reason.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-09-22 (Actual); Primary Completion 2018-02-19 (Actual); Study Completion 2018-02-19 (Actual)

PRIMARY OUTCOMES:
5-HT6 Receptor Occupancy (RO) | Treatment day 10 (24 hours post dose)
  RO in the region of interest will be calculated as 100 × (1 - BPND(treatment) / BPND(baseline)) where BPND is the binding potential
Idalopirdine plasma concentration (CPET) | Prior to and after PET scan on treatment day 10
  CPET is the concentration at the time of PET scan, defined as (CprePET + CpostPET) / 2 (average of the pre- and post-PET scanning measurements).

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — H. Lundbeck A/S
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States